CLINICAL TRIAL: NCT01455428
Title: An 8-week Randomized, Double Blind, Multi-center, Placebo-controlled Study To Evaluate The Efficacy, Safety And Tolerability Of Pregabalin ( 300mg/Day ) Using A Fixed Dosing Schedule In The Treatment Of Subjects With Postherpetic Neuralgia ( Phn )
Brief Title: Pregabalin for Treatment of Patients With Postherpetic Neuralgia (PHN)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Pfizer's Upjohn has merged with Mylan to form Viatris Inc. (Industry)
Responsible Party: Sponsor
Organization: Pfizer (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: A0081276
Record Dates: First submitted 2011-10-17; First posted 2011-10-20 (Estimated); Results first posted 2015-05-22 (Estimated); Last update posted 2021-01-28 (Actual); Status verified 2015-05

CONDITIONS: Postherpetic Neuralgia ( PHN )
Keywords: Pregabalin; Postherpetic Neuralgia ( PHN )
MeSH Terms: conditions — Neuralgia, Postherpetic | interventions — Pregabalin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Lyrica (pregabalin) (Experimental)
  Interventions: Drug: Lyrica (pregabalin)
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Lyrica (pregabalin) — Capsule, 300 mg/d, BID, 8 weeks treatment
  Arms: Lyrica (pregabalin)
Drug: Placebo — Capsule, 300 mg/d, BID, 8 weeks treatment
  Arms: Placebo

SUMMARY:
To prove pregabalin is effective in relieving pain compared with placebo in subjects with postherpetic neuralgia (PHN).

ELIGIBILITY:
Inclusion Criteria:

* Male or female Chinese subjects, ages ≥18 at screening
* Subjects with symptoms of neuropathic pain associated with postherpetic neuralgia (PHN). Subjects must have pain present for ﹥3 months after healing of the acute herpes zoster skin rash
* At screening (V1), subjects must have a score ≥40mm on the 100-mm visual analog scale (VAS) of the Short Form-McGill Pain Questionnaire (SF-MPQ, see Appendix 3)
* At randomization (V2), subjects must have a score ≥40mm on the 100-mm visual analog scale (VAS) of the Short Form-McGill Pain Questionnaire (SF-MPQ, see Appendix 3)
* At randomization (V2), subjects must have completed at least 5 daily pain diaries (DPRS, see Appendix 2) and have an average daily pain score ≥4 over the past 7 days

Exclusion Criteria:

* Subjects who demonstrate a high response to placebo, with 30% decrease on the Pain Visual Analog Scale (VAS) at randomization as compared to screening
* Subjects who have a high variability in pain scores during the 1 week screening period, with any difference between two scores ﹥3

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 223 (Actual)
Dates: Start 2011-12; Primary Completion 2014-01 (Actual); Study Completion 2014-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (22):
- China (22):
  - Peking University First Hospital, Beijing, Beijing Municipality
  - Sun Yat-Sen Memorial Hospital, Sun Yat-Sen University, Guangzhou, Guangdong
  - Shenzhen People's Hospital, Shenzhen, Guangdong
  - Union Hospital of Tongji Medical College, Huazhong University of Science and Technology, Wuhan, Hubei
  - Tongji Hospital Tongji Medical College, Huazhong University of Science and Technology, Wuhan, Hubei
  - Neurology Department, Jiangsu Province Hospital, Nanjing, Jiangsu
  - The Second Affiliated Hospital of Soochow University/Neurology Department, Suzhou, Jiangsu
  - Qilu Hospital of Shandong University, Jinan, Shandong
  - The First Affiliated Hospital of College of Medicine, Zhejiang University/Dermatology and STD Dept., Hangzhou, Zhejiang
  - Sir Run Run Shaw Hospital Affiliated of College of Medicine, Zhejiang University/Neurology Dept., Hangzhou, Zhejiang
  - Beijing Friendship Hospital, Capital Medical University/Department of Internal Neurology, Beijing
  - Peking University Third Hospital, Neurology Department, Beijing
  - Neurology Department, Beijing Hospital of the Ministry of Health, Beijing
  - West China Hospital of Sichuan University, Neurology Department, Chengdu/wuhou D
  - the first affiliated hospital ,chongqing medical university, Department of Neurology, Chongqing
  - GuangZhou First Municipal People's Hospital, Guangzhou
  - The Third Affiliated Hospital of Sun Yat-sen University, Guangzhou
  - Neurology Department, Shanghai Changzheng Hospital, Shanghai
  - Ruijin Hospital Affiliated to Shanghai Jiaotong University School of Medicine, Shanghai
  - Huashan Hospital, Fudan University/Neurology Department, Shanghai
  - Renji Hospital Shanghai Jiao Tong University School of Medicine/Neurology Department, Shanghai
  - Tianjin Medical University General Hospital, Dermatological Department, Tianjin

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A0081276&StudyName=Pregabalin%20for%20Treatment%20of%20Patients%20with%20Postherpetic%20Neuralgia%20%28PHN%29%20

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 223 participants were randomized, as stated on clinicaltrials.gov. However, 1 was randomized by mistake, was considered a screen failure, and was not given any medication. As such, the actual number of participants randomized and assigned to treatment was 222.
Groups:
- Pregabalin: Participants received 1 matching placebo capsule twice a day (BID) for 1 week (run-in period), followed by an 8-week double-blind treatment phase (1-week dose-titration phase where participants received pregabalin 150 milligram [mg] per day in the form of 75 mg BID and a 7-week fixed dose phase where participants received pregabalin 300 mg per day in the form of 150 mg BID), and a 1-week taper-off phase where participants received pregabalin 150 mg per day (in the form of 75 mg BID).
- Placebo: Participants received matching placebo capsule(s) for a period of 10 weeks.
Period: Overall Study
Arm/Group | Pregabalin | Placebo
Started | 112 | 110
Treated | 111 | 109
Completed | 98 | 92
Not Completed | 14 | 18
Not completed — Protocol Violation | 2 | 1
Not completed — Adverse Event | 6 | 2
Not completed — Lost to Follow-up | 1 | 1
Not completed — Withdrawal by Subject | 2 | 5
Not completed — Did not meet entrance criteria | 0 | 2
Not completed — Insufficient clinical response | 0 | 2
Not completed — Did not receive treatment | 1 | 1
Not completed — Other | 2 | 4

BASELINE CHARACTERISTICS:
Population: All randomized and treated participants were included in the baseline characteristics summarization.
Groups:
- Total: Total of all reporting groups
Arm/Group | Pregabalin | Placebo | Total
Number analyzed (Participants) | 111 | 109 | 220
Age, Customized [Number; unit: participants]
  18-44 years | 4 | 3 | 7
  45-64 years | 39 | 47 | 86
  More than or equal to (>=)65 years | 68 | 59 | 127
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 54 | 47 | 101
  Male | 57 | 62 | 119

OUTCOME MEASURES:

1. Primary Outcome: Baseline Mean Pain Score
Description: The daily pain rating scale (DPRS) consists of an 11-point numeric scale ranging from 0 (no pain) to 10 (worst possible pain). Participants described their pain during the past 24 hours by choosing the appropriate number between 0 and 10.
Time Frame: Baseline
Population: All participants in the Full Analysis Set (FAS) population (all participants randomized to treatment that received at least 1 dose of study medication) who had available data for this outcome measure. The Last Observation Carried Forward (LOCF) method was used.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Pregabalin | Placebo
Number analyzed (Participants) | 111 | 108
units on a scale | 5.93 (1.304) | 6.08 (1.266)

2. Primary Outcome: Change From Baseline in Mean Pain Score at Endpoint
Description: The daily pain rating scale (DPRS) consists of an 11-point numeric scale ranging from 0 ("no pain") to 10 ("worst possible pain"). Participants described their pain during the past 24 hours by choosing the appropriate number between 0 and 10. The mean endpoint pain score was obtained from the last 7 available DPRS scores of the daily pain diary while the participant was on study medication, up to and including the day after the last Week 8 (Day 57) dose.
Time Frame: Baseline until end of fixed dose phase (Day 57/Week 8)/Early Termination (Study Endpoint)
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Pregabalin | Placebo
Number analyzed (Participants) | 111 | 108
units on a scale | -1.81 (0.137) | -1.09 (0.142)
Statistical Analysis 1: Comparison: Pregabalin vs Placebo; Analysis performed using a general linear model with treatment and center as factors, and baseline value as a covariate; Test type: Superiority or Other; p = 0.0002, ANCOVA — Primary analysis was two-sided and performed at the 0.05 significance level; Least Squares Mean Difference = -0.71, 95% CI 2-sided [-1.08 to -0.34], Standard Error of Mean 0.188

3. Secondary Outcome: Change From Baseline in Weekly Mean Pain Score at Weeks 1 to 8
Description: The DPRS consists of an 11-point numeric scale ranging from 0 ("no pain") to 10 ("worst possible pain"). Participants described their pain during the past 24 hours by choosing the appropriate number between 0 and 10. The weekly mean pain score was the sum of the daily scores divided by the number of diary entries during that week.
Time Frame: Baseline and weekly from Weeks 1 to 8
Population: The FAS population consisted of all participants randomized to treatment that received at least 1 dose of study medication.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Pregabalin | Placebo
Number analyzed (Participants) | 111 | 109
units on a scale
  Week 1 change from baseline | -0.62 (0.108) | -0.12 (0.111)
  Week 2 change from baseline | -1.00 (0.109) | -0.35 (0.112)
  Week 3 change from baseline | -1.23 (0.109) | -0.65 (0.112)
  Week 4 change from baseline | -1.36 (0.110) | -0.85 (0.114)
  Week 5 change from baseline | -1.50 (0.110) | -0.99 (0.114)
  Week 6 change from baseline | -1.70 (0.110) | -1.11 (0.114)
  Week 7 change from baseline | -1.78 (0.111) | -1.07 (0.114)
  Week 8 change from baseline | -1.91 (0.111) | -1.21 (0.114)
Statistical Analysis 1: Comparison: Pregabalin vs Placebo; Week 1 Modelled Results. The model used was a linear mixed model with treatment, week, center, and treatment by week interaction as factors, and the baseline value as a covariate. A compound symmetry covariance structure is specified; Test type: Superiority or Other; p = 0.0010, Mixed Model Repeated Measures Analysis — All analyses were 2-sided and performed at the 0.05 significance level; Least Squares Mean Difference = -0.49, 95% CI 2-sided [-0.79 to -0.20], Standard Error of Mean 0.149
Statistical Analysis 2: Comparison: Pregabalin vs Placebo; Week 2 Modelled Results. The model used was a linear mixed model with treatment, week, center, and treatment by week interaction as factors, and the baseline value as a covariate. A compound symmetry covariance structure is specified; Test type: Superiority or Other; p < 0.0001, Mixed Model Repeated Measures Analysis — All analyses were 2-sided and performed at the 0.05 significance level; Least Squares Mean Difference = -0.65, 95% CI 2-sided [-0.94 to -0.35], Standard Error of Mean 0.150
Statistical Analysis 3: Comparison: Pregabalin vs Placebo; Week 3 Modelled Results. The model used was a linear mixed model with treatment, week, center, and treatment by week interaction as factors, and the baseline value as a covariate. A compound symmetry covariance structure is specified; Test type: Superiority or Other; p = 0.0001, Mixed Model Repeated Measures Analysis — All analyses were 2-sided and performed at the 0.05 significance level; Least Squares Mean Difference = -0.58, 95% CI 2-sided [-0.88 to -0.29], Standard Error of Mean 0.151
Statistical Analysis 4: Comparison: Pregabalin vs Placebo; Week 4 Modelled Results. The model used was a linear mixed model with treatment, week, center, and treatment by week interaction as factors, and the baseline value as a covariate. A compound symmetry covariance structure is specified; Test type: Superiority or Other; p = 0.0009, Mixed Model Repeated Measures Analysis — All analyses were 2-sided and performed at the 0.05 significance level; Least Squares Mean Difference = -0.51, 95% CI 2-sided [-0.81 to -0.21], Standard Error of Mean 0.152
Statistical Analysis 5: Comparison: Pregabalin vs Placebo; Week 5 Modelled Results. The model used was a linear mixed model with treatment, week, center, and treatment by week interaction as factors, and the baseline value as a covariate. A compound symmetry covariance structure is specified; Test type: Superiority or Other; p = 0.0009, Mixed Model Repeated Measures Analysis — All analyses were 2-sided and performed at the 0.05 significance level; Least Squares Mean Difference = -0.51, 95% CI 2-sided [-0.81 to -0.21], Standard Error of Mean 0.153
Statistical Analysis 6: Comparison: Pregabalin vs Placebo; Week 6 Modelled Results. The model used was a linear mixed model with treatment, week, center, and treatment by week interaction as factors, and the baseline value as a covariate. A compound symmetry covariance structure is specified; Test type: Superiority or Other; p = 0.0001, Mixed Model Repeated Measures Analysis — All analyses were 2-sided and performed at the 0.05 significance level; Least Squares Mean Difference = -0.59, 95% CI 2-sided [-0.89 to -0.29], Standard Error of Mean 0.153
Statistical Analysis 7: Comparison: Pregabalin vs Placebo; Week 7 Modelled Results. The model used was a linear mixed model with treatment, week, center, and treatment by week interaction as factors, and the baseline value as a covariate. A compound symmetry covariance structure is specified; Test type: Superiority or Other; p < 0.0001, Mixed Model Repeated Measures Analysis — All analyses were 2-sided and performed at the 0.05 significance level; Least Squares Mean Difference = -0.71, 95% CI 2-sided [-1.01 to -0.41], Standard Error of Mean 0.154
Statistical Analysis 8: Comparison: Pregabalin vs Placebo; Week 8 Modelled Results. The model used was a linear mixed model with treatment, week, center, and treatment by week interaction as factors, and the baseline value as a covariate. A compound symmetry covariance structure is specified; Test type: Superiority or Other; p < 0.0001, Mixed Model Repeated Measures Analysis — All analyses were 2-sided and performed at the 0.05 significance level; Least Squares Mean Difference = -0.70, 95% CI 2-sided [-1.00 to -0.40], Standard Error of Mean 0.154

4. Secondary Outcome: Baseline Mean Sleep Interference Score
Description: Pain-related sleep interference was assessed on an 11-point numerical rating scale ranging from 0 (did not interfere with sleep) to 10 (completely interfered [unable to sleep due to pain]). Participants were to describe how their pain had interfered with their sleep during the past 24 hours by choosing the appropriate number between 0 and 10.
Time Frame: Baseline
Population: All participants in the FAS population (all participants randomized to treatment that received at least 1 dose of study medication) who had available data for this outcome measure. The LOCF method was used.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Pregabalin | Placebo
Number analyzed (Participants) | 111 | 108
units on a scale | 3.81 (2.436) | 4.54 (2.027)

5. Secondary Outcome: Change From Baseline in Mean Sleep Interference Score at Endpoint
Description: Pain-related sleep interference was assessed on an 11-point numerical rating scale ranging from 0 (did not interfere with sleep) to 10 (completely interfered [unable to sleep due to pain]). Participants were to describe how their pain had interfered with their sleep during the past 24 hours by choosing the appropriate number between 0 and 10. The mean endpoint score was obtained from the last 7 available scores of the daily diary while the participant was on study medication, up to and including the day after the last Week 8 (Day 57) dose.
Time Frame: Baseline until end of fixed dose phase (Day 57/Week 8)/Early Termination (Study Endpoint)
Population: as for outcome 4
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Pregabalin | Placebo
Number analyzed (Participants) | 111 | 108
units on a scale | -1.24 (0.145) | -0.70 (0.150)
Statistical Analysis 1: Comparison: Pregabalin vs Placebo; Analysis performed using a general linear model with treatment and center as factors, and baseline value as a covariate; Test type: Superiority or Other; p = 0.0079, ANCOVA — Analysis was two-sided and performed at the 0.05 significance level; Least Squares Mean Difference = -0.54, 95% CI 2-sided [-0.93 to -0.14], Standard Error of Mean 0.200

6. Secondary Outcome: Change From Baseline in Weekly Mean Sleep Interference Scores at Weeks 1 to 8
Description: Pain-related sleep interference was assessed on an 11-point numerical rating scale ranging from 0 (did not interfere with sleep) to 10 (completely interfered [unable to sleep due to pain]). Participants were to describe how their pain had interfered with their sleep during the past 24 hours by choosing the appropriate number between 0 and 10. The weekly mean score was the sum of the daily scores divided by the number of diary entries during that week.
Time Frame: Baseline and weekly from Weeks 1 to 8
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Pregabalin | Placebo
Number analyzed (Participants) | 111 | 109
units on a scale
  Week 1 change from baseline | -0.52 (0.124) | 0.01 (0.128)
  Week 2 change from baseline | -0.82 (0.124) | -0.16 (0.128)
  Week 3 change from baseline | -0.92 (0.125) | -0.35 (0.129)
  Week 4 change from baseline | -0.96 (0.125) | -0.51 (0.130)
  Week 5 change from baseline | -1.02 (0.126) | -0.62 (0.130)
  Week 6 change from baseline | -1.13 (0.126) | -0.74 (0.130)
  Week 7 change from baseline | -1.27 (0.126) | -0.79 (0.130)
  Week 8 change from baseline | -1.31 (0.126) | -0.84 (0.131)
Statistical Analysis 1: Comparison: Pregabalin vs Placebo; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p = 0.0024, Mixed Model Repeated Measures Analysis — Analysis was two-sided and performed at the 0.05 significance level; Least Squares Mean Difference = -0.52, 95% CI 2-sided [-0.86 to -0.19], Standard Error of Mean 0.172
Statistical Analysis 2: Comparison: Pregabalin vs Placebo; [analysis description as in outcome 3, analysis 2]; Test type: Superiority or Other; p = 0.0002, Mixed Model Repeated Measures Analysis — Analysis was two-sided and performed at the 0.05 significance level; Least Squares Mean Difference = -0.65, 95% CI 2-sided [-0.99 to -0.31], Standard Error of Mean 0.173
Statistical Analysis 3: Comparison: Pregabalin vs Placebo; [analysis description as in outcome 3, analysis 3]; Test type: Superiority or Other; p = 0.0012, Mixed Model Repeated Measures Analysis — Analysis was two-sided and performed at the 0.05 significance level; Least Squares Mean Difference = -0.57, 95% CI 2-sided [-0.91 to -0.22], Standard Error of Mean 0.173
Statistical Analysis 4: Comparison: Pregabalin vs Placebo; [analysis description as in outcome 3, analysis 4]; Test type: Superiority or Other; p = 0.0101, Mixed Model Repeated Measures Analysis — Analysis was two-sided and performed at the 0.05 significance level; Least Squares Mean Difference = -0.45, 95% CI 2-sided [-0.79 to -0.11], Standard Error of Mean 0.174
Statistical Analysis 5: Comparison: Pregabalin vs Placebo; [analysis description as in outcome 3, analysis 5]; Test type: Superiority or Other; p = 0.0258, Mixed Model Repeated Measures Analysis — Analysis was two-sided and performed at the 0.05 significance level; Least Squares Mean Difference = -0.39, 95% CI 2-sided [-0.73 to -0.05], Standard Error of Mean 0.175
Statistical Analysis 6: Comparison: Pregabalin vs Placebo; [analysis description as in outcome 3, analysis 6]; Test type: Superiority or Other; p = 0.0260, Mixed Model Repeated Measures Analysis — Analysis was two-sided and performed at the 0.05 significance level; Least Squares Mean Difference = -0.39, 95% CI 2-sided [-0.74 to -0.05], Standard Error of Mean 0.175
Statistical Analysis 7: Comparison: Pregabalin vs Placebo; [analysis description as in outcome 3, analysis 7]; Test type: Superiority or Other; p = 0.0062, Mixed Model Repeated Measures Analysis — Analysis was two-sided and performed at the 0.05 significance level; Least Squares Mean Difference = -0.48, 95% CI 2-sided [-0.83 to -0.14], Standard Error of Mean 0.175
Statistical Analysis 8: Comparison: Pregabalin vs Placebo; [analysis description as in outcome 3, analysis 8]; Test type: Superiority or Other; p = 0.0081, Mixed Model Repeated Measures Analysis — Analysis was two-sided and performed at the 0.05 significance level; Least Squares Mean Difference = -0.47, 95% CI 2-sided [-0.81 to -0.12], Standard Error of Mean 0.176

7. Secondary Outcome: Percentage of 30 Percent (%) Responders at Endpoint
Description: The DPRS consists of an 11-point numeric scale ranging from 0 ("no pain") to 10 ("worst possible pain"). Participants described their pain during the past 24 hours by choosing the appropriate number between 0 and 10. A 30% responder was a participant who had 30% reduction or more in mean pain score at the end of the fixed dose phase (Day 57/Week 8)/Early Termination (Study Endpoint) compared to baseline.
Time Frame: End of fixed dose phase (Day 57/Week 8)/Early Termination (Study Endpoint)
Population: as for outcome 4
Measure: Number; unit: percentage of participants
Arm/Group | Pregabalin | Placebo
Number analyzed (Participants) | 111 | 108
percentage of participants | 52.3 [42.6 to 61.8] | 30.6 [22.1 to 40.2]
Statistical Analysis 1: Comparison: Pregabalin vs Placebo; Cochran-Mantel-Haenszel test comparing pregabalin to placebo adjusted for center; Test type: Superiority or Other; p = 0.0007, Cochran-Mantel-Haenszel — Analysis was two-sided and performed at the 0.05 significance level

8. Secondary Outcome: Change From Baseline in Short Form McGill Pain Questionnaire (SF-MPQ) Score at Weeks 1, 3, 5, and 8
Description: SF-MPQ was assessed according to the participant's answer to the SF-MPQ questionnaire. The score for each composite scale (sensory, affective, and total) was derived by summing the reported intensity value for each item within a particular scale where None=0, Mild=1, Moderate=2, and Severe=3. The sensory score was the sum of the scores of the first 11 pain descriptors (throbbing, shooting, stabbing, sharp, cramping, gnawing, hot-burning, aching, heavy, tender, and splitting) and could range from 0-33. The affective score was the sum of the scores of the last 4 pain descriptors (tiring-exhausting, sickening, fearful, and punishing-cruel) and could range from 0-12. The total score was the sum of the scores of all 15 pain descriptors and could range from 0 to 45. Higher scores indicated greater pain.
Time Frame: Baseline; Weeks 1, 3, 5, and 8
Population: The FAS population consisted of all participants randomized to treatment that received at least 1 dose of study medication. N=the number of participants who were evaluable for this measure at the given time point.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Pregabalin | Placebo
Number analyzed (Participants) | 111 | 109
units on a scale
  Sensory score, Baseline | 8.24 (5.276) | 8.00 (4.939)
  Sensory score, Week 1 change (N=111, 106) | -1.68 (3.776) | -0.29 (3.009)
  Sensory score, Week 3 change (N=107, 101) | -2.97 (3.852) | -1.05 (3.810)
  Sensory score, Week 5 change (N=102, 96) | -3.31 (4.496) | -1.79 (4.058)
  Sensory score, Week 8 change (N=98, 93) | -3.61 (4.299) | -1.94 (4.418)
  Affective score, Baseline | 1.25 (2.038) | 1.31 (2.124)
  Affective score, Week 1 change (N=111, 105) | -0.61 (1.602) | -0.28 (1.404)
  Affective score, Week 3 change (N=107, 100) | -0.80 (1.772) | -0.46 (1.507)
  Affective score, Week 5 change (N=102, 95) | -0.85 (2.036) | -0.59 (1.512)
  Affective score, Week 8 change (N=97,90) | -0.96 (1.941) | -0.66 (1.630)
  Total score, Baseline | 9.50 (6.621) | 9.29 (6.465)
  Total score, Week 1 change (N=111, 106) | -2.29 (4.486) | -0.57 (3.494)
  Total score, Week 3 change (N=107, 101) | -3.77 (4.761) | -1.51 (4.654)
  Total score, Week 5 change (N=102, 96) | -4.17 (5.632) | -2.37 (5.035)
  Total score, Week 8 change (N=98, 93) | -4.57 (5.117) | -2.53 (5.308)

9. Secondary Outcome: Baseline Pain Visual Analogue Scale (VAS) and Present Pain Intensity (PPI) Scale
Description: The VAS was part of the Short Form McGill Pain Questionnaire (SF-MPQ) scale and reflected the overall pain intensity score, The pain VAS was a horizontal line; 100 millimeters (mm) in length, was self-administered by the participant in order to rate pain from 0 (no pain) to 100 (worst possible pain). The PPI was part of the SF-MPQ scale and measured the participant's present pain intensity on a 6-point scale ranging from 0 (no pain) to 5 (excruciating).
Time Frame: Baseline
Population: The FAS population consisted of all participants randomized to treatment that received at least 1 dose of study medication. The LOCF method was used in the analysis of this outcome measure. Number of participants evaluable for PPI=110, 108
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Pregabalin | Placebo
Number analyzed (Participants) | 111 | 109
units on a scale
  VAS | 60.39 (13.064) | 62.60 (12.252)
  PPI | 2.33 (0.940) | 2.42 (0.738)

10. Secondary Outcome: Change From Baseline in Pain VAS From the SF-MPQ at Endpoint
Description: The VAS was part of the SF-MPQ scale and reflected the overall pain intensity score. The pain VAS was a horizontal line; 100 mm in length, was self-administered by the participant in order to rate pain from 0 (no pain) to 100 (worst possible pain).
Time Frame: Baseline to Day 57 (Week 8)/Early Termination (Study Endpoint)
Population: as for outcome 4
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Pregabalin | Placebo
Number analyzed (Participants) | 110 | 106
units on a scale | -20.71 (1.412) | -12.53 (1.451)
Statistical Analysis 1: Comparison: Pregabalin vs Placebo; Analysis performed using a general linear model with treatment and center as factors, and baseline value as a covariate; Test type: Superiority or Other; p < 0.0001, ANCOVA — Analysis was two-sided and performed at the 0.05 significance level; Least Squares Mean Difference = -8.18, 95% CI 2-sided [-11.99 to -4.37], Standard Error of Mean 1.932

11. Secondary Outcome: Change From Baseline in PPI Scale From the SF-MPQ at Endpoint
Description: The PPI was part of the SF-MPQ scale and measured the participant's present pain intensity on a 6-point scale ranging from 0 (no pain) to 5 (excruciating).
Time Frame: Baseline to Day 57 (Week 8)/Early Termination (Study Endpoint)
Population: as for outcome 4
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Pregabalin | Placebo
Number analyzed (Participants) | 110 | 105
units on a scale | -0.79 (0.078) | -0.42 (0.080)
Statistical Analysis 1: Comparison: Pregabalin vs Placebo; Analysis performed using a general linear model with treatment and center as factors, and baseline value as a covariate; Test type: Superiority or Other; p = 0.0007, ANCOVA — Analysis was two-sided and performed at the 0.05 significance level; Least Squares Mean Difference = -0.37, 95% CI 2-sided [-0.58 to -0.16], Standard Error of Mean 0.107

12. Secondary Outcome: Baseline Medical Outcomes Study (MOS)-Sleep Scale Scores
Description: The MOS-Sleep Scale was a participant-rated questionnaire consisting of 12 items that assessed key constructs of sleep. Instrument scoring yielded 7 subscales (sleep disturbance, snoring, awaken short of breath or with a headache, quantity of sleep, optimal sleep, sleep adequacy, and somnolence) as well as a 9-item overall sleep problems index. The total score ranged from 0 to 100. With the exception of sleep adequacy, optimal sleep, and quantity, higher scores reflected greater impairment in the MOS-Sleep subscales. The MOS-Sleep Scale was used to evaluate sleep during the previous week.
Time Frame: Baseline
Population: The FAS population consisted of all participants randomized to treatment that received at least 1 dose of study medication. The LOCF method was used in the analysis of this outcome measure.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Pregabalin | Placebo
Number analyzed (Participants) | 111 | 109
units on a scale
  Sleep disturbance score | 36.09 (25.542) | 35.08 (22.365)
  Snoring score | 29.19 (32.450) | 30.83 (35.017)
  Awaken short of breath score | 9.91 (21.213) | 8.07 (18.282)
  Quantity of sleep score | 6.05 (1.534) | 5.97 (1.524)
  Sleep adequacy score | 57.66 (31.449) | 60.46 (29.008)
  Somnolence score | 32.25 (19.950) | 30.89 (17.816)
  Sleep problems index score | 31.38 (20.691) | 29.27 (17.292)

13. Secondary Outcome: Change From Baseline in MOS-Sleep Scale, Sleep Disturbance Score at Endpoint
Description: The MOS-Sleep Scale was a participant-rated questionnaire consisting of 12 items that assessed key constructs of sleep. Instrument scoring yielded 7 subscales (sleep disturbance, snoring, awaken short of breath or with a headache, quantity of sleep, optimal sleep, sleep adequacy, and somnolence) as well as a 9-item overall sleep problems index. The total score ranged from 0 to 100. For sleep disturbance, the subscale score also ranged from 0 to 100, with higher scores representing greater sleep disturbance.
Time Frame: Baseline and Day 57 (Week 8)/Early Termination (Study Endpoint)
Population: All participants in the FAS population (all participants randomized to treatment that received at least 1 dose of study medication) who had available data for this outcome measure.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Pregabalin | Placebo
Number analyzed (Participants) | 103 | 97
units on a scale | -11.97 (1.821) | -4.76 (1.871)
Statistical Analysis 1: Comparison: Pregabalin vs Placebo; Analysis performed using a general linear model with treatment and center as factors, and baseline value as a covariate; Test type: Superiority or Other; p = 0.0039, ANCOVA — Analysis was two-sided and performed at the 0.05 significance level; Least Squares Mean Difference = -7.21, 95% CI 2-sided [-12.08 to -2.35], Standard Error of Mean 2.464

14. Secondary Outcome: Change From Baseline in MOS-Sleep Scale, Snoring Score at Endpoint
Description: The MOS-Sleep Scale was a participant-rated questionnaire consisting of 12 items that assessed key constructs of sleep. Instrument scoring yielded 7 subscales (sleep disturbance, snoring, awaken short of breath or with a headache, quantity of sleep, optimal sleep, sleep adequacy, and somnolence) as well as a 9-item overall sleep problems index. The total score ranged from 0 to 100. The snoring subscale score also ranged from 0 to 100, with lower scores indicating less snoring.
Time Frame: Baseline and Day 57 (Week 8)/Early Termination (Study Endpoint)
Population: as for outcome 13
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Pregabalin | Placebo
Number analyzed (Participants) | 104 | 97
units on a scale | -2.00 (2.043) | -3.73 (2.131)
Statistical Analysis 1: Comparison: Pregabalin vs Placebo; Analysis performed using a general linear model with treatment and center as factors, and baseline value as a covariate; Test type: Superiority or Other; p = 0.5351, ANCOVA — Analysis was two-sided and performed at the 0.05 significance level; Least Squares Mean Difference = 1.73, 95% CI 2-sided [-3.76 to 7.22], Standard Error of Mean 2.783

15. Secondary Outcome: Change From Baseline in MOS-Sleep Scale, Awaken Short of Breath Score at Endpoint
Description: The MOS-Sleep Scale was a participant-rated questionnaire consisting of 12 items that assessed key constructs of sleep. Instrument scoring yielded 7 subscales (sleep disturbance, snoring, awaken short of breath or with a headache, quantity of sleep, optimal sleep, sleep adequacy, and somnolence) as well as a 9-item overall sleep problems index. The total score ranged from 0 to 100. The awaken short of breath subscale also ranged from 0 to 100, with lower scores indicating less difficulty in breathing.
Time Frame: Baseline and Day 57 (Week 8)/Early Termination (Study Endpoint)
Population: as for outcome 13
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Pregabalin | Placebo
Number analyzed (Participants) | 104 | 96
units on a scale | -0.10 (1.895) | 0.26 (1.988)
Statistical Analysis 1: Comparison: Pregabalin vs Placebo; Analysis performed using a general linear model with treatment and center as factors, and baseline value as a covariate; Test type: Superiority or Other; p = 0.8892, ANCOVA — Analysis was two-sided and performed at the 0.05 significance level; Least Squares Mean Difference = -0.36, 95% CI 2-sided [-5.45 to 4.73], Standard Error of Mean 2.579

16. Secondary Outcome: Change From Baseline in MOS-Sleep Scale, Quantity of Sleep Score at Endpoint
Description: The MOS-Sleep Scale was a participant-rated questionnaire consisting of 12 items that assessed key constructs of sleep. Instrument scoring yielded 7 subscales (sleep disturbance, snoring, awaken short of breath or with a headache, quantity of sleep, optimal sleep, sleep adequacy, and somnolence) as well as a 9-item overall sleep problems index. The total score ranged from 0 to 100. The MOS Sleep Quantity sub-scale scores ranged from 0 to 24 (number of hours slept).
Time Frame: Baseline and Day 57 (Week 8)/Early Termination (Study Endpoint)
Population: as for outcome 13
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Pregabalin | Placebo
Number analyzed (Participants) | 101 | 96
units on a scale | 0.69 (0.108) | 0.25 (0.111)
Statistical Analysis 1: Comparison: Pregabalin vs Placebo; Analysis performed using a general linear model with treatment and center as factors, and baseline value as a covariate; Test type: Superiority or Other; p = 0.0035, ANCOVA — Analysis was two-sided and performed at the 0.05 significance level; Least Squares Mean Difference = 0.43, 95% CI 2-sided [0.14 to 0.72], Standard Error of Mean 0.147

17. Secondary Outcome: Percentage of Participants Who Had Optimal Sleep at Endpoint
Description: The MOS-Sleep Scale was a participant-rated questionnaire consisting of 12 items that assessed key constructs of sleep. Instrument scoring yielded 7 subscales (sleep disturbance, snoring, awaken short of breath or with a headache, quantity of sleep, optimal sleep, sleep adequacy, and somnolence) as well as a 9-item overall sleep problems index. The total score ranged from 0 to 100. The MOS optimal sleep subscale was a binary outcome derived from the sleep quantity responses: the response was YES if sleep quantity was 7 or 8 hours per night.
Time Frame: Day 57 (Week 8)/Early Termination (Study Endpoint)
Population: All participants in the FAS population (consisted of all participants randomized to treatment that received at least 1 dose of study medication) with available data to contribute to the analysis.
Measure: Number; unit: percentage of participants
Arm/Group | Pregabalin | Placebo
Number analyzed (Participants) | 101 | 96
percentage of participants | 49.5 [39.4 to 59.6] | 40.6 [30.7 to 51.1]
Statistical Analysis 1: Comparison: Pregabalin vs Placebo; Analysis performed using a logistic regression model with treatment and center as factors, and baseline value as a covariate; Test type: Superiority or Other; p = 0.0972, Regression, Logistic — Analysis was two-sided and performed at the 0.05 significance level; Odds Ratio (OR) = 1.80, 95% CI 2-sided [0.90 to 3.60]

18. Secondary Outcome: Change From Baseline in MOS-Sleep Scale, Sleep Adequacy Score at Endpoint
Description: The MOS-Sleep Scale was a participant-rated questionnaire consisting of 12 items that assessed key constructs of sleep. Instrument scoring yielded 7 subscales (sleep disturbance, snoring, awaken short of breath or with a headache, quantity of sleep, optimal sleep, sleep adequacy, and somnolence) as well as a 9-item overall sleep problems index. The total score ranged from 0 to 100. The sleep adequacy subscale also ranged from 0 to 100, with higher scores indicating greater sleep adequacy.
Time Frame: Baseline and Day 57 (Week 8)/Early Termination (Study Endpoint)
Population: as for outcome 13
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Pregabalin | Placebo
Number analyzed (Participants) | 103 | 97
units on a scale | 10.44 (2.325) | 8.64 (2.403)
Statistical Analysis 1: Comparison: Pregabalin vs Placebo; Analysis performed using a general linear model with treatment and center as factors, and baseline value as a covariate; Test type: Superiority or Other; p = 0.5702, ANCOVA — Analysis was two-sided and performed at the 0.05 significance level; Least Squares Mean Difference = 1.80, 95% CI 2-sided [-4.44 to 8.03], Standard Error of Mean 3.161

19. Secondary Outcome: Change From Baseline in MOS-Sleep Scale, Somnolence Score at Endpoint
Description: The MOS-Sleep Scale was a participant-rated questionnaire consisting of 12 items that assessed key constructs of sleep. Instrument scoring yielded 7 subscales (sleep disturbance, snoring, awaken short of breath or with a headache, quantity of sleep, optimal sleep, sleep adequacy, and somnolence) as well as a 9-item overall sleep problems index. The total score ranged from 0 to 100. The somnolence subscale score also ranged from 0 to 100, with lower scores indicating less somnolence.
Time Frame: Baseline and Day 57 (Week 8)/Early Termination (Study Endpoint)
Population: as for outcome 13
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Pregabalin | Placebo
Number analyzed (Participants) | 104 | 97
units on a scale | 0.33 (1.613) | -0.54 (1.668)
Statistical Analysis 1: Comparison: Pregabalin vs Placebo; Analysis performed using a general linear model with treatment and center as factors, and baseline value as a covariate; Test type: Superiority or Other; p = 0.6929, ANCOVA — Analysis was two-sided and performed at the 0.05 significance level; Least Squares Mean Difference = 0.87, 95% CI 2-sided [-3.46 to 5.20], Standard Error of Mean 2.194

20. Secondary Outcome: Change From Baseline in MOS-Sleep Scale, Sleep Problems Index Score at Endpoint
Description: The MOS-Sleep Scale was a participant-rated questionnaire consisting of 12 items that assessed key constructs of sleep. Instrument scoring yielded 7 subscales (sleep disturbance, snoring, awaken short of breath or with a headache, quantity of sleep, optimal sleep, sleep adequacy, and somnolence) as well as a 9-item overall sleep problems index. The total score ranged from 0 to 100. The sleep problems index subscale score also ranged from 0 to 100, with lower scores indicating fewer sleep problems.
Time Frame: Baseline and Day 57 (Week 8)/Early Termination (Study Endpoint)
Population: as for outcome 13
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Pregabalin | Placebo
Number analyzed (Participants) | 102 | 96
units on a scale | -7.38 (1.427) | -4.54 (1.471)
Statistical Analysis 1: Comparison: Pregabalin vs Placebo; Analysis performed using a general linear model with treatment and center as factors, and baseline value as a covariate; Test type: Superiority or Other; p = 0.1403, ANCOVA — Analysis was two-sided and performed at the 0.05 significance level; Least Squares Mean Difference = -2.84, 95% CI 2-sided [-6.63 to 0.94], Standard Error of Mean 1.920

21. Secondary Outcome: Clinical Global Impression of Change (CGIC) Score at Endpoint
Description: The CGIC was a clinician-rated global measure that provided a clinically relevant and easy to interpret account of a clinician's perception of the clinical importance of the participant's improvement or worsening during their involvement in a clinical study. Clinicians rated the participant's overall improvement on a 7-point scale where scores ranged from 1 (very much improved) to 7 (very much worse).
Time Frame: Day 57 (Week 8)/Early Termination (Study Endpoint)
Population: as for outcome 13
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Pregabalin | Placebo
Number analyzed (Participants) | 104 | 97
units on a scale | 2.55 (0.086) | 3.18 (0.090)
Statistical Analysis 1: Comparison: Pregabalin vs Placebo; Analysis was performed using a general linear model with treatment and center as factors; Test type: Superiority or Other; p < 0.0001, ANOVA — Analysis was two-sided and performed at the 0.05 significance level; Least Squares Mean Difference = -0.62, 95% CI 2-sided [-0.86 to -0.39], Standard Error of Mean 0.118

22. Secondary Outcome: Patient Global Impression of Change (PGIC) Score at Endpoint
Description: The PGIC was a participant-rated global measure that provided a clinically relevant and easy to interpret account of a participant's perception of the clinical importance of their own improvement or worsening during their involvement in a clinical study. Participants rated their overall improvement on a 7-point scale where scores ranged from 1 (very much improved) to 7 (very much worse).
Time Frame: Day 57 (Week 8)/Early Termination (Study Endpoint)
Population: as for outcome 13
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Pregabalin | Placebo
Number analyzed (Participants) | 104 | 97
units on a scale | 2.68 (0.083) | 3.17 (0.086)
Statistical Analysis 1: Comparison: Pregabalin vs Placebo; Analysis was performed using a general linear model with treatment and center as factors; Test type: Superiority or Other; p < 0.0001, ANOVA — Analysis was two-sided and performed at the 0.05 significance level; Least Squares Mean Difference = -0.49, 95% CI 2-sided [-0.72 to -0.27], Standard Error of Mean 0.113

23. Secondary Outcome: Baseline Hospital Anxiety and Depression Scale (HADS) Scores
Description: The HADS was a self-administered questionnaire that consisted of 2 subscales, 1 measuring anxiety (HADS-A Scale) and the other measuring depression (HADS-D Scale). Each subscale comprised of 7 items; participants assessed how each item applied to them on a scale of 0 (no presence of anxiety or depression) to 3 (severe feeling of anxiety or depression). Subscores from HADS-A (Anxiety) and HADS-D (Depression) were not to be combined. The interpretation of each HADS subscales was as follows: 0-7 normal, 8-10 mild, 11-14 moderate and 15-21 severe.
Time Frame: Baseline
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Pregabalin | Placebo
Number analyzed (Participants) | 111 | 109
units on a scale
  Anxiety total score | 3.22 (3.921) | 3.37 (3.466)
  Depression total score | 3.45 (3.963) | 3.47 (3.387)

24. Secondary Outcome: Change From Baseline in HADS Anxiety Total Score at Endpoint
Description: The HADS was a self-administered questionnaire that consisted of 2 subscales, 1 measuring anxiety (HADS-A Scale) and the other measuring depression (HADS-D Scale). Each subscale was comprised of 7 items; participants assessed how each item applied to them on a scale of 0 (no presence of anxiety or depression) to 3 (severe feeling of anxiety or depression). Subscores from HADS-A (Anxiety) and HADS-D (Depression) were not to be combined. The interpretation of each HADS subscales was as follows: 0-7 normal, 8-10 mild, 11-14 moderate and 15-21 severe.
Time Frame: Baseline and Day 57 (Week 8)/Early Termination (Study Endpoint)
Population: as for outcome 13
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Pregabalin | Placebo
Number analyzed (Participants) | 104 | 97
units on a scale | -0.92 (0.233) | -0.71 (0.241)
Statistical Analysis 1: Comparison: Pregabalin vs Placebo; Analysis was performed using a general linear model with treatment and center as factors, and the baseline value as a covariate; Test type: Superiority or Other; p = 0.5060, ANCOVA — Analysis was two-sided and performed at the 0.05 significance level; Least Squares Mean Difference = -0.21, 95% CI 2-sided [-0.83 to 0.41], Standard Error of Mean 0.315

25. Secondary Outcome: Change From Baseline in HADS Depression Total Score at Endpoint
Description: as for outcome 24
Time Frame: Baseline and Day 57 (Week 8)/Early Termination (Study Endpoint)
Population: as for outcome 13
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Pregabalin | Placebo
Number analyzed (Participants) | 104 | 97
units on a scale | -0.65 (0.209) | -0.55 (0.217)
Statistical Analysis 1: Comparison: Pregabalin vs Placebo; [analysis description as in outcome 24, analysis 1]; Test type: Superiority or Other; p = 0.7247, ANCOVA — Analysis was two-sided and performed at the 0.05 significance level; Least Squares Mean Difference = -0.10, 95% CI 2-sided [-0.66 to 0.46], Standard Error of Mean 0.285

ADVERSE EVENTS:
Description: The same event may appear as both an AE and a SAE. However, what is presented are distinct events. An event may be categorized as serious in one participant and as nonserious in another, or one participant may have experienced both a serious and nonserious event during the study. All treated participants were included in the analysis.
Arm/Group | Pregabalin | Placebo
Serious Adverse Events (participants affected / at risk) | 2/111 | 0/109
Other Adverse Events (participants affected / at risk) | 40/111 | 21/109
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Pregabalin (N=111) | Placebo (N=109)
Respiratory tract infection (Infections and infestations) | 1 | 0
Cerebral ischaemia (Nervous system disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Pregabalin (N=111) | Placebo (N=109)
Dry mouth (Gastrointestinal disorders) | 6 | 3
Oedema peripheral (General disorders) | 7 | 2
Nasopharyngitis (Infections and infestations) | 5 | 9
Dizziness (Nervous system disorders) | 27 | 4
Somnolence (Nervous system disorders) | 6 | 5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.